CLINICAL TRIAL: NCT04335292
Title: Osimertinib Then Chemotherapy in EGFR-mutated Lung Cancer with Osimertinib Third-line Rechallenge
Acronym: OCELOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mark Vincent (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Mark Vincent, Medical Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCELOT
Record Dates: First submitted 2020-03-06; First posted 2020-04-06 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Epidermal Growth Factor Receptor Mutation; Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): First-line treatment = osimertinib, 80 mg, oral, daily; Second-line treatment = platinum (carboplatin or cisplatin) + pemetrexed chemotherapy, prescribed as per institutional standards; Third-line treatment = osimertinib rechallenge, 80 mg, oral, daily.
  Patients may enter the study at first-line treatment, second-line treatment, or third-line treatment. This is dependent on meeting the eligibility criteria.
  Interventions: Drug: Osimertinib First-Line; Drug: Platinum + Pemetrexed Chemotherapy Second-Line; Drug: Osimertinib Third-Line

INTERVENTIONS:
Drug: Osimertinib First-Line — Osimertinib, 80 mg, oral, daily
Drug: Platinum + Pemetrexed Chemotherapy Second-Line — Platinum-based chemotherapy (carboplatin or cisplatin) and pemetrexed are prescribed as per institutional standards.
Drug: Osimertinib Third-Line — Rechallenge with osimertinib, 80 mg, oral, daily

SUMMARY:
This phase II single-armed study will examine the clinical utility of retreating patients with osimertinib, in the third-line, following first-line treatment with osimertinib and second-line treatment with platinum and pemetrexed chemotherapy. The current standard of care for first-line Epidermal Growth Factor Receptor (EGFR) mutated Advanced Non-Small Cell Lung Cancer (aNSCLC) is osimertinib, followed by cytotoxic chemotherapy.

The repeat of osimertinib following previous treatment failure is investigational, although supported by scientific rationale. The dosing and scheduling of osimertinib follows its use in approved settings. The investigators examine its tolerability and efficacy in this setting to ensure osimertinib is a safe third-line option for patients with Epidermal Growth Factor Receptor mutated (EGFR+) Advanced Non-Small Cell Lung Cancer(aNSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male or female patients of at least 18 years of age
* Pathologically proven advanced non-small cell lung cancer (i.e. stage M1 (metastasis), or earlier stages if unfit or unsuitable for radical treatment). Patients must have a tissue diagnosis of lung cancer, either by histology or cytology, however, in the event that there is insufficient tissue for molecular analysis, mutations identified in circulating tumor deoxyribonucleic acid (ctDNA) analysis will be permitted.
* Patients must have a known activating Epidermal Growth Factor Receptor (EGFR) mutation. Atypical Epidermal Growth Factor Receptor (EGRF) mutations are allowed. Atypical mutations may require sponsor approval. Exon 20 insertions will not be allowed.
* Patients must have an Eastern Cooperative Oncology Group/World Health Organisation Performance Status (ECOG/WHO-PS) of 0-3 and an expectation that they could potentially receive second-line chemotherapy
* Patients must have an expected life expectancy of at least 12 weeks
* Female subjects should be using highly effective contraceptive measures, and must have a negative pregnancy test and not be breast-feeding prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
  * Women under 50 years old are consider postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) levels in the post-menopausal range for the institution
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
* Male subjects should be willing to use barrier contraception
* Additional Criteria for patients enrolling after first-line progression and prior to second-line chemotherapy::
* Subjects must have complete baseline demographic data available (age at diagnosis of metastatic non-small cell lung cancer, ethnicity, smoking status, sex, history of brain metastasis) and the following must be available (if applicable):

  o Date of first dose of osimertinib, date that first-line osimertinib was permanently discontinued, date of first-line progression.
* Additional Criteria for patients enrolling at the time of third-line osimertinib rechallenge:
* Subjects must have complete baseline demographic data available (age at diagnosis of metastatic non-small cell lung cancer (NSCLC), ethnicity, smoking status, sex, history of brain metastasis) and the following must be available (if applicable):

  o Date of first dose of osimertinib, date that first-line osimertinib was permanently discontinued, date of first-line progression, date second-line chemotherapy was started, which platinum chemotherapy was given, if pemetrexed maintenance was given, date that second-line chemotherapy was permanently stopped, and date of progression on second-line treatment.
* Patients must have received platinum/ pemetrexed chemotherapy in the second-line chemotherapy
* Subjects must have measurable disease defined as at least one measurable lesion that can be accurately assessed by Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) at baseline and follow up visits.Subjects must have measurable disease defined as at least one measurable lesion that can be accurately assessed by Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) at baseline and follow up visits.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or involved staff at the study site).
* A second invasive malignancy in the previous three years, other than localized non-melanoma skin cancer, which might be confused with the Epidermal Growth Factor Receptor (EGFR) mutated lung cancer.
* Any other serious and uncontrolled medical or psychiatric condition which would likely interfere in the conduct of the study.
* Pregnancy or lactation
* Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
* Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of Cytochrome P450 3A4 (CYP3A4) (at least 3 weeks prior). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on Cytochrome P450 3A4 (CYP3A4).
* Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2, prior platinum-therapy-related neuropathy.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Patients with spinal cord compression, symptomatic and unstable brain metastases except for those patients who have completed definitive therapy and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
* Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* Inadequate bone marrow reserve or organ function (as demonstrated by any of the following laboratory values: absolute neutrophil count less than1.5 x 10 to the power of 9/L, platelet count less than 100 x 10 to the power of 9/L, haemoglobin less than 90 g/L), alanine aminotransferase greater than 2.5 times upper limit of normal (ULN) if no demonstrable liver metastases or greater than 5 times ULN in the presence of liver metastases; aspartate aminotransferase greater than 2.5 times ULN if no demonstrable liver metastases or greater than 5 times ULN in the presence of liver metastases; total bilirubin greater than 1.5 times ULN if no liver metastases or greater than 3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases; serum creatinine greater than 1.5 times ULN concurrent with creatinine clearance less than 50 mL/min [measured or calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is greater than 1.5 times ULN.
* History of hypersensitivity to any of the active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Previous adjuvant cytotoxic chemotherapy within the 6 months prior to enrollment.
* Previous adjuvant anti programmed cell death protein 1(anti-PD-1) or anti programmed death-ligand 1 (anti-PD-L1) therapy within 90 days prior to enrollment.
* For patients enrolling prior to first-line treatment with osimertinib:
* Any previous systemic therapy for Epidermal Growth Factor Receptor mutated (EGFR+) advanced Non-Small Cell Lung Cancer (aNSCLC).
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) greater than 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
  * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities [including serum/plasma potassium less than the Lower Limit of Normal (LLN), serum/plasma magnesium greater than the Lower Limit of Normal (LLN), serum/plasma calcium less than the Lower Limit of Normal (LLN)], congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
* For patients enrolling after progression on first-line osimertinib and prior to second-line chemotherapy all patients must have:
* Received osimertinib in the first-line and no other systemic therapy for their Epidermal Growth Factor Receptor mutated (EGFR+) Advanced Non-Small Cell Lung Cancer (aNSCLC).
* For patients enrolling at the time of third-line osimertinib rechallenge all patients must have:
* Received osimertinib in the first-line followed by second-line platinum (carboplatin/cisplatin) with pemetrexed (pemetrexed maintenance is permitted), and no other systemic therapy for their Epidermal Growth Factor Receptor mutated (EGFR+) advanced Non-Small Cell Lung Cancer.
* Received a minimum of 1 dose of platinum (carboplatin/cisplatin) with pemetrexed.

  * AND
* At least 90 days have lapsed since the last dose of first-line osimertinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate according to Response Evaluation Criteria in Solid Tumors version 1.1 | End of study (approximately 4 years)
  Objective Response Rate will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Objective Response Rate is the percent of subjects with measurable disease with at least one visit response of complete response or partial response.

SECONDARY OUTCOMES:
Progression Free Survival according to Response Evaluation Criteria in Solid Tumors version 1.1 | End of study (approximately 4 years)
  Progression Free Survival will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Progression Free Survival is the time from the first dose of osimertinib until the date of objective disease progression or death (by any cause in the absence of progression).
Duration of Response according to Response Evaluation Criteria in Solid Tumors version 1.1 | End of study (approximately 4 years)
  Duration of Response will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Duration of Response is the time from the date of first documented response until date of documented progression or death (in the absence of disease progression), in the third-line setting (osimertinib re-challenge).
Disease Control Rate according to Response Evaluation Criteria in Solid Tumors version 1.1 | End of study (approximately 4 years)
  Disease Control Rate will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Disease Control Rate is the percentage of subjects who have a best overall response of complete response or partial response or stable disease.
Tumor Shrinkage according to Response Evaluation Criteria in Solid Tumors version 1.1 | End of study (approximately 4 years)
  Tumor Shrinkage will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).
Overall Survival | End of study (approximately 4 years)
  Overall Survival is the time from the date of the first osimertinib dose rechallenge (third line setting), until death due to any cause.
Time to Treatment Failure | End of study (approximately 4 years)
  Time to Treatment Failure is the time from first dose of osimertinib rechallenge (third-line setting), until the date of objective disease progression leading to the decision to proceed with the next line of systemic therapy, or permanently forego antineoplastic system therapy, or death (by any cause in the absence of progression).
Effect of Osimertinib Rechallenge on Health Related Quality of Life Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-C30 | End of study (approximately 4 years)
  The effects of osimertinib on health related quality of life will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30).
  The EORTC QLQ-C30 is a questionnaire consisting of 30 items measuring subjects general cancer symptoms and functioning. Responses regarding function and symptoms are on a scale of 1 (not at all) to 4 (very much). Also included are questions about overall health and quality of life. Responses are on a scale of 1 (very poor) to 7 (excellent).
Effect of Osimertinib Rechallenge on Health Related Quality of Life Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-LC 13 | End of study (approximately 4 years)
  The effects of osimertinib on health related quality of life will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13).
  The EORTC QLQ-LC13 is a complementary questionnaire to the EORTC QLQ-C30, measuring lung cancer symptoms. Responses regarding symptoms are on a scale of 1 (not at all) to 4 (very much).
Effect of Osimertinib Rechallenge on Disease-Related Symptoms Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaires EORTC QLQ-C30 | End of study (approximately 4 years)
  The effects of osimertinib on disease-related symptoms will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30).
  The EORTC QLQ-C30 is a questionnaire consisting of 30 items measuring subjects general cancer symptoms and functioning. Responses regarding function and symptoms are on a scale of 1 (not at all) to 4 (very much). Also included are questions about overall health and quality of life. Responses are on a scale of 1 (very poor) to 7 (excellent).
Effect of Osimertinib Rechallenge on Disease-Related Symptoms Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-LC 13 | End of study (approximately 4 years)
  The effects of osimertinib on disease-related symptoms will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer 13 items (EORTC QLQ-LC13).
  The EORTC QLQ-LC13 is a complementary questionnaire to the EORTC QLQ-C30, measuring lung cancer symptoms. Responses regarding symptoms are on a scale of 1 (not at all) to 4 (very much).
Objective Response Rate in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Objective Response Rate in the atypical Epidermal Growth Factor Receptor (EGFR) mutation population will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), in both the first line and third line settings. Objective Response Rate is the percent of subjects with measurable disease with at least one visit response of complete response or partial response.
Progression Free Survival according to Response Evaluation Criteria in Solid Tumors in the Atypical Epidermal Growth Factor Receptor Population | End of study (approximately 4 years)
  Progression Free Survival in the atypical Epidermal Growth Factor Receptor (EGFR) population will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), in both the first line and third line settings. Progression Free Survival is the time from the first dose of osimertinib until the date of objective disease progression or death (by any cause in the absence of progression).
Duration of Response according to Response Evaluation Criteria in Solid Tumors version 1.1 in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Duration of Response in the atypical Epidermal Growth Factor Receptor (EGFR) population will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), in both the first line and third line settings. Duration of Response is the time from the date of first documented response until date of documented progression or death (in the absence of disease progression), in the third-line setting (osimertinib re-challenge).
Disease Control Rate according to Response Evaluation Criteria in Solid Tumors version 1.1 in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Disease Control Rate in the atypical Epidermal Growth Factor Receptor (EGFR) population will be determined using investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), in both the first line and third line settings. Disease Control Rate is the percentage of subjects who have a best overall response of complete response or partial response or stable disease.
Tumor Shrinkage according to Response Evaluation Criteria in Solid Tumors version 1.1 in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Time to Treatment Failure is the time from first dose of osimertinib, until the date of objective disease progression leading to the decision to proceed with the next line of systemic therapy, or permanently forego antineoplastic system therapy, or death (by any cause in the absence of progression). Time to treatment failure will be analyzed in the atypical Epidermal Growth Factor Receptor (EGFR) mutation population, in both the first line and third line settings.
Overall Survival in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Overall Survival is the time from the date of the first osimertinib dose, until death due to any cause. Overall Survival will be analyzed in the atypical Epidermal Growth Factor Receptor (EGFR) mutation population, in both the first line and third line settings.
Time to Treatment Failure in the Atypical Epidermal Growth Factor Receptor Mutation Population | End of study (approximately 4 years)
  Time to Treatment Failure is the time from first dose of osimertinib, until the date of objective disease progression leading to the decision to proceed with the next line of systemic therapy, or permanently forego antineoplastic system therapy, or death (by any cause in the absence of progression). Time to Treatment Failure will be analyzed in the atypical Epidermal Growth Factor Receptor (EGFR) mutation population, in both the first line and third line settings.

OTHER OUTCOMES:
Analysis of Mutations in Circulating Tumor Deoxyribonucleic Acid Blood Samples | End of study (approximately 4 years)
  Retrospective/real-time analysis of EGFR (and other) mutations in Circulating Tumor Deoxyribonucleic acid (ctDNA) from all study subjects.
Effects of Duration on Osimertinib on Post Progression Outcomes During First-Line Treatment | End of study (approximately 4 years)
  A comparison of the effects of duration on osimertinib during first-line treatment on post progression outcomes.
Effects of Duration on Osimertinib on Post Progression Outcomes During Third-Line Treatment | End of study (approximately 4 years)
  A comparison of the effects of duration on osimertinib during third-line treatment on post progression outcomes. This includes time from first rechallenge (third-line) dose of osimertinib until subsequent treatments, and progression free survival of subsequent treatments.
Effects of Duration on Chemotherapy on Post Progression Outcomes | End of study (approximately 4 years)
  A comparison of the effects of duration on chemotherapy (second-line treatment) on post progression outcomes.
Assessment of Tumor markers and Circulating Tumor Deoxyribonucleic Acid Levels for Predictors of Radiographic Response | End of study (approximately 4 years)
  Changes to blood-based biomarkers will be analyzed and compared to objective response rate and disease control rate to see if there are predictors or associations with radiographic response.
Analysis of Genetic Markers in Blood Samples | End of study (approximately 4 years)
  Optional blood samples will be collected at various timepoints for analysis of key genetic markers.
Analysis of Genetic Markers in Tissue | End of study (approximately 4 years)
  Optional tumor samples will be collected at various timepoints for analysis of key genetic markers.
Analysis of Proteomic Markers in Blood Samples | End of study (approximately 4 years)
  Optional blood samples will be collected at various timepoints for analysis of key proteomic markers.
Analysis of Proteomic Markers in Tissue | End of study (approximately 4 years)
  Optional tumor samples and blood samples will be collected at various timepoints for analysis of key proteomic markers.
Molecular Analysis of Serial Biopsies | End of study (approximately 4 years)
  Optional serial biopsies will be collected at various timepoints and analyzed via molecular diagnostics for genetic alterations, and for the co-mutational context. Samples will be compared to Circulating Tumor Deoxyribonucleic Acid (ctDNA) samples.
Safety and Tolerability Profile of Osimertinib: Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) | End of study (approximately 4 years)
  Adverse events will be graded using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Vincent, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (10):
- Canada (10):
  - BC Cancer Agency, Vancouver, British Columbia
  - Lions Gate Hospital, Vancouver, British Columbia
  - William Osler Health System, Brampton, Ontario
  - Hamilton Health Sciences Centre, Juravinski Cancer Centre, Hamilton, Ontario
  - Grand River Regional Cancer Centre, Kitchener, Ontario
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - Durham Regional Cancer Centre, Lakeridge Health, Oshawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No